CLINICAL TRIAL: NCT06649695
Title: A Phase II Trial of Teclistamab in Participants With Previously Treated Immunoglobulin Light-chain (AL) Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Janssen Research & Development (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN40/64007957AMY2002
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: AL Amyloidosis
Keywords: teclistamab
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Teclistamab (Experimental): Teclistamab will be administered via a subcutaneous injection (SC)
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered via a subcutaneous injection (SC)
  Other Names: JNJ-64007957

SUMMARY:
This is a multicenter open-label, phase 2 study in participant with previously treated immunoglobulin light-chain (AL) Amyloidosis to evaluate the benefit of teclistamab

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of AL amyloidosis and typed with immunohistochemistry/ immunofluorescence, immunoelectron microscopy, or mass spectrometry. In patients with biopsy-confirmed amyloidosis, ambiguous amyloid typing results, and cardiac involvement alone, a negative pyrophosphate (PYP) or technetium-99m (99mTc) and 3,3-diphosphono-1,2-propanodicarboxylic acid (DPD-Tc99m) bone scan is required to distinguish cardiac involvement due to AL amyloidosis from amyloid transthyretin (ATTR) amyloidosis. Data from the initial diagnosis are accepted.
* Genetic testing must be negative for transthyretin mutations associated with hereditary amyloidosis, or immunohistochemistry/ immunofluorescence/ immunoelectron microscopy/ mass spectrometry of amyloid deposits must provide clear evidence of κ or λ light chains in patients who present with peripheral neuropathy or heart as the dominant organ involvement. Data from the initial diagnosis are accepted.
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1 or 2
* Mayo stage I-IIIA cardiac disease at Screening
* Relapsed patients must have received at least 1 line of treatment, including Dara and bortezomib. Patients must have received at least two cycles of therapy. However, patients who have received high-dose therapy with melphalan as their only therapy are also eligible.
* Measurable hematologic disease: a dFLC >20 mg/L with an abnormal κ/λ ratio (with Freelite® test kits, The Binding Site) or presence of a monoclonal spike ≥0.5 g/dL.
* Adequate bone marrow function, without transfusion or growth factors within 5 days prior to the first drug intake (C1D1), defined as:
* Absolute neutrophils ≥1,000/mm3,
* Platelets ≥75,000/mm3,
* Hemoglobin ≥8.5 g/dL.
* Adequate organ function, defined as:
* Serum creatinine clearance (CKD-EPI formula) ≥20 mL/min,
* Serum SGPT/ALT <5.0 x Upper Limit of Normal (ULN),
* Serum total bilirubin <2.0 mg/dL or direct bilirubin ≤30% of the total, unless the patient has Gilbert's syndrome, where direct bilirubin should then be <2.0 mg/dL,
* Serum albumin ≥<2.5 gr/dl (medication to correct serum albumin levels is permitted).

Exclusion Criteria:

* Amyloid-specific syndrome, such as carpal tunnel syndrome or skin purpura, as the only evidence of disease. The finding of isolated vascular amyloid in a bone marrow biopsy specimen or in a plasmacytoma is not indicative of systemic amyloidosis.
* Isolated soft-tissue involvement.
* Presence of non-AL amyloidosis.
* Previous anti-BCMA targeted therapy (including, but not limited to, bispecifics).
* Intolerance to dexamethasone that would prohibit treatment with trial therapy.
* MM diagnosed as per the International Myeloma Working Group (IMWG) criteria, with the exception of monoclonal gammopathy of unknown significance (MGUS) or smoldering Myeloma, not requiring treatment.

Note: A MM diagnosis with a serum FLC ratio >100, as the only myeloma-defining event, does NOT constitute an exclusion.

* All hematologic malignancies, with the exception of low-risk Philadelphia chromosome negative (Ph-) myeloproliferative neoplasms (MPNs) and low-risk myelodysplastic syndromes (MDS), not requiring treatment.
* Mayo stage IIIB cardiac disease at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Hematologic Complete Response (CR) rate | baseline up to 3 cycles of treatment (approximately 3 months)
  Percentage of participants achieving CR or better according to EHA/ISA guidelines

SECONDARY OUTCOMES:
Hematologic Overall Response Rate (ORR) rate | Baseline up to progression of disease or death (approximately 3,5 years)
  Percentage of participants achieving Complete Response (CR), Very Good Partial Response (VGPR) or Partial Response (PR) or better according to EHA/ISA guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Murielle Roussel, MD, Principal Investigator — CHU Limoges
Locations (10):
- Australia (2):
  - South Australia Health, Adelaide
  - Westmead Hospital, Sydney
- France (2):
  - CHU Limoges, Limoges
  - Paris St Louis, Paris
- Germany (3):
  - University Hospital Essen, Essen
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Würzburg, Würzburg
- General Hospital of Athens "Alexandra", Athens, Greece
- Fondazione I.R.C.C.S Policlinico "San Matteo", Pavia, Italy
- UMC Utrecht, Utrecht, Netherlands